CLINICAL TRIAL: NCT04414423
Title: Combination of Bone Marrow Concentrate and Iliac Cancellous Bone Graft in Alveolar Cleft Grafting: a Clinical & Radiographic Evaluation
Brief Title: Combination of Bone Marrow Concentrate and Iliac Cancellous Bone Graft in Alveolar Cleft Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Alshaimaa Ahmed shabaan, associate professor in oral & maxillofacial Surgery Department, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMC AlvCleft
Record Dates: First submitted 2020-05-25; First posted 2020-06-04 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Alveolar Cleft Grafting
Keywords: bone marrow concentrate; alveolar cleft; CBCT; Bone density; bone volume

STUDY DESIGN:
Intervention Model Description: Eighteen patients will be divided into two equal groups. Each group comprises nine patients.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bone marrow concentrate (Experimental): Bone marrow concentrate combined with Autogenous bone graft
  Interventions: Procedure: bone marrow concentrate alveolar cleft grafting
- autogenous bone graft (Active Comparator): grafting with autogenous bone graft
  Interventions: Procedure: Autogenous alveolar grafting

INTERVENTIONS:
Procedure: bone marrow concentrate alveolar cleft grafting — patients will undergo surgery to repair alveolar cleft with autogenous bone graft combined with bone marrow concentrate
  Arms: Bone marrow concentrate
Procedure: Autogenous alveolar grafting — patients will undergo surgery to repair alveolar cleft with autogenous bone graft
  Arms: autogenous bone graft

SUMMARY:
The aim of this study will be to analyze the newly formed bone volume and density, 6 months after alveolar cleft grafting using iliac cancellous bone graft, with and without bone marrow concentrate.

DETAILED DESCRIPTION:
Twelve patients with unilateral alveolar cleft will be enrolled in this randomized comparative study.

The patients will be divided into two groups, the control (group A) who received illiac cancellous bone graft and study group who received a combination of bone marrow concentrate and illiac cancellous bone graft (group B).

Cone Beam CT (CBCT) images will be done prior to surgery to asses preoperative alveolar defect volume. Six months postoperative CBCT images will be done and postoperative newly bone formed volume and density will be evaluated and bone formation ratio (BF%) will be calculated as follows: BF% = (formed volume/alveolar defect) × 100%.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from maxillary alveolar cleft
* Patient with Primary, complete cleft lip

Exclusion Criteria:

* Syndromic cases will be excluded
* Previous operated cases

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
bone volume | six months postoperative
  V= (A1xT) + ( A2 xT) + …….+ (An xT) where: V= volume A= area T= thickness of the axial C.T slice N=number of slices

SECONDARY OUTCOMES:
bone density | six months postoperative
  the average bone density will be measured from the CBCT
bone formation ratio | six months postoperative
  BF% = (formed volume/alveolar defect) × 100%.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Dentistry, Al Fayyum
  - Faculty of Dentistry, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pinheiro FHSL, Drummond RJ, Frota CM, Bartzela TN, Dos Santos PB. Comparison of early and conventional autogenous secondary alveolar bone graft in children with cleft lip and palate: A systematic review. Orthod Craniofac Res. 2020 Nov;23(4):385-397. doi: 10.1111/ocr.12394. Epub 2020 Jun 28. PMID 32446283
- [Background] Ziegler CG, Van Sloun R, Gonzalez S, Whitney KE, DePhillipo NN, Kennedy MI, Dornan GJ, Evans TA, Huard J, LaPrade RF. Characterization of Growth Factors, Cytokines, and Chemokines in Bone Marrow Concentrate and Platelet-Rich Plasma: A Prospective Analysis. Am J Sports Med. 2019 Jul;47(9):2174-2187. doi: 10.1177/0363546519832003. Epub 2019 Apr 29. PMID 31034242
- [Derived] Shabaan AA, Salahuddin A, Aboulmagd I, Ragab R, Salah KA, Rashid A, Ayad HM, El Aty Ahmed WA, Refahee SM. Alveolar cleft reconstruction using bone marrow aspirate concentrate and iliac cancellous bone: A 12-month randomized clinical study. Clin Oral Investig. 2023 Nov;27(11):6667-6675. doi: 10.1007/s00784-023-05276-9. Epub 2023 Oct 5. PMID 37794139